CLINICAL TRIAL: NCT05254873
Title: Long-term Follow-up of Patients Included in the EYE-TAR(MA) Study: Rehabilitation of Facial Emotion Recognition in Alzheimer's Disease and Study of the Consequences on Gaze Strategy, Behavior Disorders and Family Caregivers' Burden
Brief Title: Long-term Follow-up of Patients Included in the EYE-TAR(MA) Study.
Status: Completed | Type: Observational
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: EYE-TAR(MA)-FU
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer's Dementia (AD); Family Caregivers
Keywords: Video-oculography; Eye-Tracking; Gaze strategies; Training of Affect Recognition; Emotion recognition; Behavioral disorders; Caregiver's burden; Alzheimer's Dementia; Oculomotor behaviors; Facial emotion recognition
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AD-TAR: AD subjects who took part to Facial Emotion Recognition rehabilitation (TAR) during EYE-TAR(MA) study
  Interventions: Other: Long term follow-up
- AD-Cognitive Stim: AD subjects who took part to cognitive stimulation session (12 sessions during 4 weeks) during EYE-TAR(MA) study
  Interventions: Other: Long term follow-up

INTERVENTIONS:
Other: Long term follow-up — Long term follow-up for patient who completed the EYE-TAR(MA) study.

SUMMARY:
EYE-TAR(MA)-Follow-Up is a non-interventionel, long-term follow-up study in subjects who participated to the study referred as EYE-TAR(MA) (NCT04730440)

EYE-TAR(MA)-Follow-Up aims to evaluate the long-term impacts of the Training of Affect Recognition TAR (an emotion recognition rehabilitation program), on social cognition abilities, evolve gaze strategies, behavioral disorders, and the caregiver's burden in Alzheimer's disease (AD).

Subjects who completed EYE-TAR(MA) study, and who have signed informed consent for this follow-up, will be eligible to enroll. They will attend one visit two years post EYE-TAR(MA) study intervention (intervention was TAR, or a "classic" cognitive stimulation program) to undergo the following evaluation: Eye-tracking recording during Ekman Faces task, Mini Mental State Examination (MMSE), Neuropsychiatric Inventory (NPI), Zarit scale (completed by caregiver).

DETAILED DESCRIPTION:
It is commonly admitted that social cognition impairment, like deficit in facial emotion recognition or misinterpretation of others' intentions (Theory of Mind), are associated with social behavior disorders.

This kind of disorders are observed in Fronto-Temporal Dementia (FTD), Alzheimer's Dementia (AD) and Parkinson's Disease (PD), with severe deficits in FTD and lighter deficits in AD and PD. One explanation is that patients apply inappropriate visual exploration strategies to decode emotions and intentions of others.

The study EYE-TAR(MA), NCT04730440, aimed to evaluate impacts of an emotion recognition rehabilitation program, named Training of Affect Recognition (TAR), on social cognition abilities (facial emotion recognition and theory of mind) in AD. In addition, investigators hypothesized that the effect of this rehabilitation will also evolve gaze strategies, behavioral disorders, and the caregiver's burden.

EYE-TAR(MA) results showed that participants who participated to the TAR (a) recognized facial emotions better and faster, especially sadness, fear and neutral expression; (b) evolved their gaze strategies on emotional faces with increased observation of the upper part of the face (nose and / or eyes); (c) had reduced behavioral disorders and the caregiver's burden. These results were specific to the TAR, since no significant change was observed in the AD-Control group who had participated in a "classic" cognitive stimulation program.

These changes were generally maintained one month after treatment.

Because there is not long-term follow-up data for these patients, Sponsor and investigators set-up the EYE-TAR(MA)-Follow-Up study to evaluate the long-term impacts of the Training of Affect Recognition, on social cognition abilities, evolve gaze strategies, behavioral disorders, and the caregiver's burden.

Subjects who completed EYE-TAR(MA) study, and who have signed informed consent for this follow-up, will be eligible to enroll. They will attend a visit two years post EYE-TAR(MA) study intervention to undergo the following evaluation: Eye-tracking recording during Ekman Faces task, Mini Mental State Examination (MMSE), Neuropsychiatric Inventory (NPI), Zarit scale (completed by caregiver).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were included in the EYE-TAR (MA) study, and who completed this study.
* Subject accompanied by the caregiver already present during participation in the EYE-TAR (MA) study.
* Written informed consent signed by patient and family caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AD patients, who completed EYE-TAR(MA) study, and who have signed informed consent for this 2 years follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Facial emotion recognition (FER) performances | 2 years follow-up
  Change from EYE-TAR(MA) Last evaluation and Comparison of FER performance between Long-term follow-up AD-TAR group and Long-term follow-up AD-Cognitive Stimulation group.
  Evaluation criteria: Scores to Ekman Faces task (1976) and time to answer. FER was assessed using pictures from the Ekman Faces task (1976), to test the recognition of the six facial basic emotions and neutral faces. There were four pictures per emotion, for a total of 28. For each picture, participants were asked to select one of the seven labels (anger, disgust, fear, sadness, happiness, surprise and neutral), with a maximum of 8 seconds of response time per picture.

SECONDARY OUTCOMES:
Eye gaze strategies during Facial emotion recognition (FER) | 2 years follow-up
  Change from EYE-TAR(MA) Last evaluation and Comparison of gaze patterns between Long-term follow-up AD-TAR group and Long-term follow-up AD-Cognitive Stimulation group.
  Evaluation criteria: Eye movements (number and duration of fixations on areas of interest) recorded with an eye-tracking device. FER was assessed using some pictures from the Ekman Faces task (1976).
Behavioral disorders | 2 years follow-up
  Change from EYE-TAR(MA) Last evaluation and Comparison between Long-term follow-up AD-TAR group and Long-term follow-up AD-Cognitive Stimulation group.
  Evaluation criteria: Neuropsychiatric Inventory (NPI), a scale that includes ten behavioral items (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability and aberrant motor behaviors) and two neurovegetative symptoms (sleep and appetite disorders). The evaluation was based on an interview with patients' primary caregivers. Both the frequency (/5) and the severity (/3) of each behavior were determined and a score was calculated by multiplying the frequency and the severity of each behavior observed during the last month.
The Family caregiver's burden | 2 years follow-up
  Change from EYE-TAR(MA) Last evaluation and Comparison between Long-term follow-up AD-TAR group and Long-term follow-up AD-Cognitive Stimulation group.
  Evaluation criteria: The burden of the family caregiver was measured with the Zarit scale (completed by the caregiver). Composed of 22 questions on the physical, emotional and financial load felt. Total score /88.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine LOUCHART DE LA CHAPELLE, MD-PhD, Principal Investigator — Centre Mémoire, Centre de Gérontologie Clinique RAINIER III, Princess Grace Hospital, Monaco
Locations (1):
- Centre Mémoire / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Polet K, & al. Remédiation de la reconnaissance des émotions faciales dans la maladie d'Alzheimer et effets sur les stratégies d'observation, les troubles du comportement et le fardeau de l'aidant. Neurol psychiatr gériatr, 2021 ; 21(12 — https://doi.org/10.1016/j.npg.2020.08.003
- See also: Mirzai M, & al. Long-term effects of rehabilitation of facial emotion recognition and its clinical consequences in Alzheimer's disease — https://doi.org/10.1016/j.npg.2023.03.006